CLINICAL TRIAL: NCT05804500
Title: Safety and Engagement in Cardiac Rehabilitation With the RecoveryPlus Telerehabilitation Platform: A Prospective, Single-arm, Pilot Study
Brief Title: RecoveryPlus Telerehab Platform Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NODEHealth Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro00070335
Record Dates: First submitted 2023-03-27; First posted 2023-04-07 (Actual); Last update posted 2024-01-19 (Actual); Status verified 2024-01

CONDITIONS: Heart Diseases; Angina, Stable; Angina Pectoris; Myocardial Ischemia; Myocardial Infarction; Coronary Artery Disease; Coronary Artery Stenosis; Valve Heart Disease; Valve Disease, Heart
MeSH Terms: conditions — Heart Diseases; Angina, Stable; Angina Pectoris; Myocardial Ischemia; Myocardial Infarction; Coronary Artery Disease; Coronary Stenosis; Heart Valve Diseases | interventions — Receptors, Calcitonin

STUDY DESIGN:
Intervention Model Description: In this prospective, single-arm study, we will look at the initiation, participation, sustained engagement, and safety of 100 adult subjects (ages 45 years or older) with recent (within the past 60 days) clinician referral to CR who are offered CTR via the RecoveryPlus platform.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cardiac Telerehabilitation Arm (Experimental): In this prospective, single-arm study, we will look at the initiation, participation, sustained engagement, and safety of 100 adult subjects (ages 45 years or older) with recent (within the past 60 days) clinician referral to CR who are offered CTR via the RecoveryPlus platform.
  Interventions: Behavioral: Cardiac Telerehabilitation (CTR) via the RecoveryPlus platform

INTERVENTIONS:
Behavioral: Cardiac Telerehabilitation (CTR) via the RecoveryPlus platform — RecoveryPlus has developed an innovative CTR platform for patients with CVD that leverages: (1) video conferencing functionality (Zoom) for synchronous telehealth sessions of CR instruction for patients and licensed exercise physiologists (EPs), (2) a patient-facing mobile application delivering asynchronous exercise videos, and (3) a health care provider web portal for clinicians and EPs. The RecoveryPlus platform includes the ability for EPs and clinicians to monitor patient clinical data (e.g., heart rate) and input (e.g., rating of difficulty for individual exercises) and tailor individual patient regimens regularly for increased safety and optimal outcomes.

SUMMARY:
In this prospective, single-arm study, we will look at the initiation, participation, sustained engagement, and safety of 100 adult subjects (ages 45 years or older) with recent (within the past 60 days) clinician referral to CR who are offered CTR via the RecoveryPlus platform. We want to understand the effectiveness of the RecoveryPlus platform in engaging participants in CR while remaining a safe alternative for the delivery of evidence-based CR content.

The primary hypothesis of this study is that the RecoveryPlus CTR platform and patient-facing mobile application provide a safe alternative to traditional in-person CR, and demonstrate a high rate of initiation, participation, and engagement in CR exercise programming than traditional modes of CR delivery, as documented in the literature. Current in-person and non-personalized CR programming lacks RecoveryPlus' convenient remote access, easy-to-use digital tools to support independent, autonomous exercise, and a platform to facilitate engagement and feedback between patients and EPs.

DETAILED DESCRIPTION:
1 BACKGROUND INFORMATION AND RATIONALE 1.1 Introduction Cardiac rehabilitation (CR) is an evidence-based program designed to help individuals with heart disease recover and improve their physical, psychological, and social functioning. CR is an important component in the management of patients with cardiovascular disease, which aims to reduce the risk of subsequent cardiovascular events and improve quality of life. However, traditional modes of CR delivery such as in-person sessions, have limitations, including low participation rates and inconvenience for patients. Telehealth technology may provide a viable alternative, and the RecoveryPlus platform has been developed specifically to deliver evidence-based CR content remotely.

1.2 Clinical Need Cardiovascular diseases (CVDs) are the leading cause of morbidity and mortality worldwide, and their incidence and prevalence have steadily risen over the past decades. Several common cardiovascular diseases include coronary heart disease, heart surgery cerebrovascular disease, rheumatic heart disease, deep vein thrombosis, congestive heart failure, and pulmonary embolism. The Million Hearts Cardiac Rehabilitation Collaborative, co-led by the Centers for Disease Control and Prevention (CDC) and the Centers for Medicare and Medicaid Services (CMS), aimed to prevent one million CVD events by 2027. However, there were only 2,300 CR programs in the U.S. in 2021.

1.3 Clinical Rationale This study will capture metrics that demonstrate the effectiveness and safety of RecoveryPlus in engaging participants in a 12-week, hybrid, synchronous/asynchronous remote CR program, thus contributing to study subjects' recovery from a precipitating cardiac health condition.

1.4 Design Rationale Given that RecoveryPlus is a remote CR platform that includes synchronous telehealth visits with a licensed Exercise Physiologist (EP) and a patient-facing mobile application offering tools for asynchronous exercise guidance, the study will be conducted entirely remotely. Study data, including clinical endpoints, will be collected per usual RecoveryPlus program participation.

1.5 Proposed Solution Safe, effective remote cardiac telerehabilitation (RCR) offers a scalable solution to the need for greater engagement of patients recovering from CVD events in evidence-based CR exercise programming. CR generally is a multi-faceted approach that combines exercise training, patient education, nutritional counseling, risk factor behavior modification (e.g., around management of lipids, blood pressure, weight, smoking) to improve outcomes of patients with CVD and reduce associated morbidity and mortality.4 In particular, physical activity has become a core component of CR programs as mortality risk is lower among patients who meet WHO recommendations for physical activity.5 Over the past decade, the use of home-based programs for CR has become more prevalent, as they expand access to rehabilitation for patients with limited mobility, and allow providers to manage a broader panel of patients.4 As with many healthcare services, the COVID-19 pandemic accelerated the transition of many CR programs to home-based care, also termed telerehabilitation or CTR.6 Status Quo: CR is a safe, effective, evidence-based intervention that remains severely underutilized by patients for a variety of reasons, including: inconvenience, lack of incorporation of patient input and capacity for personalization, and poorly designed, static content. Therefore, while proven effective, the lack of initiation and engagement of patients in CR programming means it falls short of its potential to widely impact patient outcomes.

1.6 Device Description RecoveryPlus has developed an innovative CTR platform for patients with CVD that leverages: (1) video conferencing for synchronous telehealth sessions of CR instruction for patients and licensed EPs, (2) a patient-facing mobile application delivering asynchronous exercise videos, and (3) a health care provider web portal for clinicians and EPs. The RecoveryPlus platform includes the ability for EPs and clinicians to monitor patient clinical data (e.g., heart rate) and input (e.g., rating of difficulty for individual exercises) and tailor individual patient regimens regularly for increased safety and optimal outcomes.

The main goal of RecoveryPlus is to engage and motivate patients to achieve sustained engagement in their cardiac rehabilitation in a safe environment. The RecoveryPlus team has done this by solving the problem experienced by medical professionals who otherwise lacked reliable clinical and adherence data needed to understand patients' CR experience in real-time. The solution is a purpose-built platform incorporating synchronous telehealth visits with licensed EPs along with a mobile medical application to be used for asynchronous exercise instruction. With exercise videos and personalized heart rate targets, and continuous readings during exercise sessions, RecoveryPlus provides patients with more robust instruction, monitoring, and support, and medical professionals the tools to guide patients' exercise, track patients' heart rates and receive patients' feedback. Data derived from a heart rate monitor as well as the patient's feedback is reviewed by medical professionals to assess exercise intensity, the patient's conditions, and adherence to the prescribed exercise.

Patients are asked for frequent feedback on their exercise experience. Individual exercises are followed by prompts to rate the perceived level of difficulty [1-10 scale] of the exercise. If a patient chooses to skip an exercise, the app asks the reason [too hard, cannot reach target HR, pain, personal reasons] and requires qualitative characterization of the reason before being allowed to continue. If a patient chooses to exit a session prior to completion, the app asks for a reason [uncomfortable, too tired, movement too hard, personal business] and requires qualitative characterization of the reason. Unlike current practice, the RecoveryPlus platform provides the capability for real-time, automated alerts sent to RecoveryPlus personnel for any negative symptom report or out-of-range heart rate reading and immediate evaluation to determine the severity of a symptom and what follow-up course of action is required (if any). Patients are instructed as part of regular RecoveryPlus programming practice to stop exercising and report any cardiac-related symptom to their clinician or EP at any time, during or outside of exercise sessions. RecoveryPlus staff receive and respond to alerts 24 hours/7 days per week.

The healthcare provider web portal allows clinicians and EPs to enter a patient's basic demographic and clinical information, create fitness assessments, define and update a patient's exercise prescription, provide educational information, and generate wellness reports.

ELIGIBILITY:
Inclusion Criteria:

* • Older adult [age 45+]

  * Meets criteria and receives clinician referral to CR
  * Within 60 days of referring cardiac event
  * Ambulatory
  * Under medical management and deemed stable by a clinician
  * Low to moderate risk of exercise-induced cardiac event
  * Any CR eligible diagnosis in the past 12 months as defined by Medicare Part B coverage excluding heart/heart-lung transplant. Medicare Part B covers CR for patients who experience 1 or more of the following:

    * Acute myocardial infarction within the preceding 12 months
    * Coronary artery bypass surgery
    * Current stable angina pectoris
    * Heart valve repair or replacement
    * Percutaneous transluminal coronary angioplasty or coronary stenting
    * Stable, chronic heart failure is defined as patients with left ventricular ejection fraction of 35% or less and New York Heart Association (NYHA) class II to III symptoms despite being on optimal heart failure medical therapy for at least 6 weeks.

Exclusion Criteria:

* • Body mass index (BMI) equal to or over 35

  * Hospitalization or significant decline in health between recruitment-consent and start of the study
  * Physical or mental health limitations that prohibit participation in CR exercise activities
  * Less than a basic facility with smartphone/tablet
  * Lack of access to WIFI
  * No active email address
  * Hearing and/or sight impairment that would limit the ability to follow exercise videos and instructions.
  * Non-English-speaking
  * Unable to read in English.

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2023-03-27 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-01-15 (Actual)

PRIMARY OUTCOMES:
INITIATION | 3 months
  Initiation will be defined as the proportion of enrolled screen-eligible patients who completed all baseline assessments and completed the initial CTR session.
PARTICIPATION | 3 months
  Participation will be defined as the proportion of prescribed CTR sessions per participant that are completed (51% or more of prescribed session length completed) throughout the 12-week study period.
SUSTAINED ENGAGEMENT | 3 months
  Sustained engagement will be defined as the proportion of enrolled participants who had a minimum of 1 completed session, synchronous and/or asynchronous, per week (within each 7day interval from the initial session) for at least 9 weeks of the 12-week study period.
SAFETY | 3 months
  Safety will be measured as the total number of adverse events over the entire course of the 12-week study period.

SECONDARY OUTCOMES:
6-minute WALK TEST | 3 months
  This endpoint will be defined as the difference in fitness as measured by performance on a 6-minute walk test from baseline to endline. The 6-minute walk test is a widely used and well documented measure of aerobic exercise capacity used to indicate change in fitness.7 In this test, one measures the distance an individual is able to walk over a total of six minutes on a hard flat surface. Per routine RecoveryPlus practice, the EP will instruct participants virtually on completion of the test at baseline and again at endline.
RESTING HEART RATE | 3 months
  This endpoint will be defined as the difference in fitness as measured by resting heart rate from baseline to endline. Resting heart rate is positively associated with mortality and is known to lower with regular exercise. Per routine RecoveryPlus practice, the EP will instruct participants virtually on completion of resting heart rate assessment at baseline and again at endline.
QUALITY OF LIFE | 3 months
  QoL will be defined as the difference in score on the Short-Form Health Survey (SF-36), a validated and commonly used measure of patient perceived quality of life and functional health and wellbeing, from baseline to endline.8 During the initial teleheath evaluation appointment, EPs will provide a link to a secure web form and facilitate participant completion of the baseline SF-36 online; after 12 weeks, EPs will facilitate completion of an endline SF-36 using the same process.

CONTACTS AND LOCATIONS:
Overall Officials: Nitin G Vaswani, MD, Principal Investigator — NODEHealth Foundation
Locations (1):
- NODEHealth Foundation, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No
Data collection is the responsibility of the clinical trial staff at the site under the supervision of the site PI, all based in the U.S. The investigator is responsible for ensuring the accuracy, completeness, legibility, and timeliness of the data reported. Data from the devices and subject questionnaires will be stored in a 21 CFR Part 11-compliant data capture system. The data system includes password protection and internal quality checks, such as automatic range checks, to identify data that appear inconsistent, incomplete, or inaccurate.

REFERENCES:
- [Background] Scheinowitz M, Harpaz D. Safety of cardiac rehabilitation in a medically supervised, community-based program. Cardiology. 2005;103(3):113-7. doi: 10.1159/000083433. Epub 2005 Jan 19. PMID 15665529
- [Background] Thompson PD, Franklin BA, Balady GJ, Blair SN, Corrado D, Estes NA 3rd, Fulton JE, Gordon NF, Haskell WL, Link MS, Maron BJ, Mittleman MA, Pelliccia A, Wenger NK, Willich SN, Costa F; American Heart Association Council on Nutrition, Physical Activity, and Metabolism; American Heart Association Council on Clinical Cardiology; American College of Sports Medicine. Exercise and acute cardiovascular events placing the risks into perspective: a scientific statement from the American Heart Association Council on Nutrition, Physical Activity, and Metabolism and the Council on Clinical Cardiology. Circulation. 2007 May 1;115(17):2358-68. doi: 10.1161/CIRCULATIONAHA.107.181485. PMID 17468391
- [Background] Pavy B, Iliou MC, Meurin P, Tabet JY, Corone S; Functional Evaluation and Cardiac Rehabilitation Working Group of the French Society of Cardiology. Safety of exercise training for cardiac patients: results of the French registry of complications during cardiac rehabilitation. Arch Intern Med. 2006 Nov 27;166(21):2329-34. doi: 10.1001/archinte.166.21.2329. PMID 17130385
- [Background] Thomas RJ, Beatty AL, Beckie TM, Brewer LC, Brown TM, Forman DE, Franklin BA, Keteyian SJ, Kitzman DW, Regensteiner JG, Sanderson BK, Whooley MA. Home-Based Cardiac Rehabilitation: A Scientific Statement From the American Association of Cardiovascular and Pulmonary Rehabilitation, the American Heart Association, and the American College of Cardiology. Circulation. 2019 Jul 2;140(1):e69-e89. doi: 10.1161/CIR.0000000000000663. Epub 2019 May 13. PMID 31082266
- [Background] Meinhart F, Stutz T, Sareban M, Kulnik ST, Niebauer J. Mobile Technologies to Promote Physical Activity during Cardiac Rehabilitation: A Scoping Review. Sensors (Basel). 2020 Dec 24;21(1):65. doi: 10.3390/s21010065. PMID 33374322
- [Background] Kemps HMC, Brouwers RWM, Cramer MJ, Jorstad HT, de Kluiver EP, Kraaijenhagen RA, Kuijpers PMJC, van der Linde MR, de Melker E, Rodrigo SF, Spee RF, Sunamura M, Vromen T, Wittekoek ME; Committee for Cardiovascular Prevention and Cardiac Rehabilitation of the Netherlands Society of Cardiology. Recommendations on how to provide cardiac rehabilitation services during the COVID-19 pandemic. Neth Heart J. 2020 Jul;28(7-8):387-390. doi: 10.1007/s12471-020-01474-2. PMID 32676982
- [Background] Bellet RN, Adams L, Morris NR. The 6-minute walk test in outpatient cardiac rehabilitation: validity, reliability and responsiveness--a systematic review. Physiotherapy. 2012 Dec;98(4):277-86. doi: 10.1016/j.physio.2011.11.003. Epub 2012 May 16. PMID 23122432
- [Background] Lins L, Carvalho FM. SF-36 total score as a single measure of health-related quality of life: Scoping review. SAGE Open Med. 2016 Oct 4;4:2050312116671725. doi: 10.1177/2050312116671725. eCollection 2016. PMID 27757230
- [Derived] Bilbrey T, Martin J, Zhou W, Bai C, Vaswani N, Shah R, Chokshi S, Chen X, Bhusri S, Niemi S, Meng H, Lei Z. A Dual-Modality Home-Based Cardiac Rehabilitation Program for Adults With Cardiovascular Disease: Single-Arm Remote Clinical Trial. JMIR Mhealth Uhealth. 2024 Oct 1;12:e59098. doi: 10.2196/59098. PMID 39150858